CLINICAL TRIAL: NCT02919592
Title: MemoryShape® and MemoryGel® Breast Implants Post Approval New Enrollment Study ("Glow Study")
Brief Title: Memory Gel and Shape Combined Cohort
Acronym: Glow
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEN-15-003
Record Dates: First submitted 2016-09-23; First posted 2016-09-29 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Primary Breast Augmentation; Primary Breast Reconstruction; Revision Breast Augmentation; Revision Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Primary Breast Augmentation (Experimental): Participants who meet the requirements for primary breast augmentation (have not had previous silicone or saline breast implants) and have been implanted with Mentor MemoryGel® Breast Implants or MemoryShape® Breast Implants
  Interventions: Device: MemoryShape® Breast Implants; Device: MemoryGel® Breast Implants
- Revision Breast Augmentation (Experimental): Participants who meet the requirements for revision breast augmentation (have had previous silicone or saline breast implants) and have been implanted with Mentor MemoryGel® Breast Implants or MemoryShape® Breast implants
  Interventions: Device: MemoryShape® Breast Implants; Device: MemoryGel® Breast Implants
- Primary Breast Reconstruction (Experimental): Participants who meet the requirements for primary breast reconstruction (have not had previous silicone or saline breast implants, not including tissue expanders) and have been implanted with Mentor MemoryGel® Breast Implants or MemoryShape® Breast Implants
  Interventions: Device: MemoryShape® Breast Implants; Device: MemoryGel® Breast Implants
- Revision Breast Reconstruction (Experimental): Participants who meet the requirements for revision breast reconstruction (have had previous silicone or saline breast implants) and have been implanted with Mentor MemoryGel® Breast Implants or MemoryShape® Breast Implants
  Interventions: Device: MemoryShape® Breast Implants; Device: MemoryGel® Breast Implants
- Other Aesthetic Surgery (Active Comparator): Participants who meet the requirements for other aesthetic surgery procedures, which may not include silicone implants (breast or otherwise)
  Interventions: Procedure: Other Aesthetic Surgery

INTERVENTIONS:
Device: MemoryShape® Breast Implants — MENTOR® MemoryShape™ Breast Implants are devices with shells constructed from medical grade silicone elastomer. The shell is filled with Mentor's proprietary formulation of medical grade silicone gel. The textured shell is constructed of successive crosslinked layers of silicone elastomer, and includes raised orientation marks on the anterior and posterior of the implant intended to help the physician orient the implant and ensure proper placement during implantation. Each MENTOR® MemoryShape™ Breast Implant is provided sterile. MemoryShape Breast Implants are available in sizes ranging from 120 cc-775 cc and 5 styles with various projection and height options.
  Arms: Primary Breast Augmentation; Primary Breast Reconstruction; Revision Breast Augmentation; Revision Breast Reconstruction
Device: MemoryGel® Breast Implants — MENTOR® MemoryGel™ Breast Implants are round devices with shells constructed from medical grade silicone elastomer. The shell is filled with MemoryGel™, Mentor's proprietary formulation of medical grade silicone gel, and is constructed of successive cross-linked layers of silicone elastomer. There are two styles of shell: smooth and textured. Each MENTOR® MemoryGel™ Breast Implant is provided sterile. MemoryGel Breast Implants are available in sizes ranging from 100 cc-800 cc and 4 styles with various projection and height options.
  Arms: Primary Breast Augmentation; Primary Breast Reconstruction; Revision Breast Augmentation; Revision Breast Reconstruction
Procedure: Other Aesthetic Surgery — Other aesthetic surgery procedures (for example, liposuction, rhinoplasty, brow lift, rhytidectomy, mentoplasty/genioplasty, otoplasty, or blepharoplasty; may not include silicone implants)
  Arms: Other Aesthetic Surgery

SUMMARY:
The purpose of this study is to collect additional post-approval clinical data on the long-term performance of MemoryShape and MemoryGel Breast Implants, as indicated for primary or revisional breast augmentation and primary or revisional breast reconstruction.

DETAILED DESCRIPTION:
The post-approval study will include a maximum of 3500 women undergoing breast augmentation or reconstruction with MemoryShape or MemoryGel Breast Implants. Four cohorts will be included: primary augmentation, revision-augmentation, primary reconstruction, and revision-reconstruction. For the purpose of assessing rheumatological and neurological signs and symptoms, a control group with 300-480 women will be selected from the participating investigators' practices, who are undergoing an aesthetic surgery other than breast implant surgery. Breast implant patients and the concurrent control group patients will be followed for 10 years. Baseline and operative data will be collected at the beginning of the study, and follow-up data will be collected annually for 10 years through online questionnaires.

ELIGIBILITY:
Inclusion Criteria MemoryShape and MemoryGel Breast Implant Patients (Prospectively Enrolled):

1. Is a candidate for breast augmentation with MemoryShape or MemoryGel Breast Implants and is at least 22 years old (primary or revision) OR is a candidate for breast reconstruction (primary or revision) with MemoryShape or MemoryGel Breast Implants and is at least 18 years old;
2. Signs an Acknowledgement of Informed Decision from the patient brochure, or equivalent documentation of discussion and acknowledgement;
3. Signs an Informed Consent Form, including an Authorization to Disclose Health Information and Release Medical Records;
4. Agrees to answer baseline questions;
5. Agrees to authorize return of the device(s) to Mentor if the device is explanted during study participation;
6. Agrees via Informed Consent to comply with study follow-up, including following the surgeon's standard of care for office visits and responding to questionnaires in their entirety; and
7. Has a valid e-mail address and access to the internet to complete online questionnaires.

Exclusion Criteria MemoryShape and MemoryGel Breast Implant Patients (Prospectively Enrolled):

1. Has active infection anywhere in her body;
2. For augmentation patients, has a history of cancer of any kind, except non-melanoma skin cancer; for reconstruction patients, has a history of cancer of any kind, except non melanoma skin cancer or adequately treated breast cancer;
3. Has a confirmed diagnosis of connective tissue disease or neurological disease OR is currently being evaluated for symptoms suggestive of connective tissue disease or neurological disease;
4. Is currently pregnant or nursing;
5. Is planning on undergoing or has undergone bariatric surgery; or
6. Is planning on undergoing experimental procedures or procedures with investigational products/devices during the study period that in the opinion of the investigator could compromise the results of this study.

Inclusion Criteria Concurrent Control Group (Other Aesthetic Surgery) Patients (Prospectively Enrolled):

1. Is a candidate for aesthetic surgery (for example, liposuction, rhinoplasty, brow lift, autoplasty, rhytidectomy, mentoplasty/genioplasty, otoplasty, or blepharoplasty; may not include silicone or saline implants) and is at least 22 years of age;
2. Signs an Informed Consent Form, including an Authorization to Disclose Health Information and Release Medical Records;
3. Agrees to answer baseline questions;
4. Agrees via Informed Consent to comply with study follow-up, including responding to questionnaires in their entirety; and
5. Has a valid e-mail address and access to the internet to complete online questionnaires.

Exclusion Criteria Concurrent Control Group (Other Aesthetic Surgery) Patients (Prospectively Enrolled):

1. Has ever had unilateral or bilateral breast implants (including breast tissue expanders);
2. Expects to undergo breast implant surgery during the study period;
3. Has ever had silicone implants anywhere in her body;
4. Has active infection anywhere in her body;
5. Has a history of cancer of any kind, except non-melanoma skin cancer;
6. Has a confirmed diagnosis of connective tissue disease or neurological disease OR is currently being evaluated for symptoms suggestive of connective tissue disease or neurological disease;
7. Is currently pregnant or nursing;
8. Is planning on undergoing or has undergone bariatric surgery; or
9. Is planning on undergoing experimental procedures or procedures with investigational products/devices during the study period that in the opinion of the investigator could compromise the results of this study.

Inclusion Criteria MemoryShape Breast Implant Patients (Retrospectively Enrolled):

1. Received MemoryShape Breast Implants for breast augmenation after January 01, 2015 and was at least 22 years old (primary or revision) at the time of surgery OR underwent breast reconstruction (primary or revision) with MemoryShape Breast Implants after January 01, 2015. A women who has since had her MemoryShape Breast Implants explanted may still be enrolled in the study.
2. Signed an Acknowledgement of Informed Decision from the patient brochure, or equivalent documentation of discussion and acknowledgement is available from the time of surgery;
3. Signs an Informed Consent Form, including an Authorization to Disclose Health Information and Release Medical Records;
4. Agrees to answer baseline questions;
5. Agrees to authorize return of the device(s) to Mentor if the device is explanted during study participation;
6. Agrees via Informed Consent to comply with study follow-up, including following the surgeon's standard of care for office visits and responding to questionnaires in their entirety; and
7. Has a valid e-mail address and access to the internet to complete online questionnaires.

Exclusion Criteria MemoryShape Breast Implant Patients (Retrospectively Enrolled):

1. Had an active infection anywhere in her body at the time of surgery;
2. For augmentation patients, had a history of cancer (prior to implantation) of any kind, except non-melanoma skin cancer; for reconstruction patients, had a history of cancer (prior to implantation) of any kind, except non melanoma skin cancer or adequately treated breast cancer;
3. Had a confirmed diagnosis of connective tissue disease or neurological disease prior to implantation OR was being evaluated for symptoms suggestive of connective tissue disease or neurological disease;
4. Was pregnant or nursing at the time of surgery;
5. Was planning on undergoing bariatric surgery at the time of breast implant surgery or has undergone bariatric surgery since breast implant surgery; or
6. Is planning on undergoing experimental procedures or procedures with investigational products/devices during the study period that in the opinion of the investigator could compromise the results of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3613 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2031-06-16 (Estimated); Study Completion 2031-06-16 (Estimated)

PRIMARY OUTCOMES:
10 Year Kaplan-Meier estimated cumulative incidence rate of occurrence of local complications | 10 years

SECONDARY OUTCOMES:
Rates of occurrence of connective tissue disease | 10 years
Rates of occurrence of rheumatological signs and symptoms | 10 years
Rates of occurrence of neurological signs and symptoms | 10 years
Rates of occurrence of cancer | 10 years
Rates of occurrence of suicide | 10 years
Rates of lactation complications | 10 years
Rates of MRI confirmed rupture | 10 years
Effectiveness | 10 years
  Patient satisfaction rates

OTHER OUTCOMES:
PROMIS (Patient-Reported Outcome Measures Information System) Health Measure Questionnaire for Fatigue | Baseline, 10 years
  Short Form 4a
PROMIS (Patient-Reported Outcome Measures Information System) Health Measure Questionnaire for Cognitive Function Abilities | Baseline, 10 years
  Short Form 6a

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Mentor Worldwide, LLC
Locations (78):
- United States (78):
  - Hedden Plastic Surgery Center, Birmingham, Alabama
  - Plastic Surgery of Tuscaloosa, Tuscaloosa, Alabama
  - Advanced Plastic Surgery Institute, Gilbert, Arizona
  - Advanced Surgical Associates, Mesa, Arizona
  - Robles Plastic Surgery, Phoenix, Arizona
  - Berardi Aesthetics and Plastic Surgery, Scottsdale, Arizona
  - Guerra Plastic Surgery Center, Scottsdale, Arizona
  - Mark Malek, MD Plastic Surgery, Scottsdale, Arizona
  - Vanderpool Cosmetic Plastic Surgery, Fayetteville, Arkansas
  - Jaime Schwartz, MD, Beverly Hills, California
  - Susan E. Downey, MD Inc, Burbank, California
  - Mohebali Plastic Surgery, Corte Madera, California
  - Institute of Cosmetic and Reconstructive Surgery, Fountain Valley, California
  - Newport Beach Center for Plastic Surgery, Newport Beach, California
  - Newport Center for Special Surgery, Newport Beach, California
  - North Coast Plastic Surgery, Oceanside, California
  - Li Plastic Surgery, Ontario, California
  - Summit Plastic Surgery, Redding, California
  - Verve Plastic Surgery, Solana Beach, California
  - Kaweah Delta Health Care District, Visalia, California
  - Park Meadows Cosmetic Surgery, Lone Tree, Colorado
  - David Bogue MD, Plastic Surgery, PL, Boca Raton, Florida
  - The Plastic Surgery Institute of Miami, Coral Gables, Florida
  - University of Miami / Sylvester Comp Cancer Ctr, Coral Gables, Florida
  - South Florida Plastic Surgery, Fort Lauderdale, Florida
  - First Coast Plastic Surgery, Jacksonville, Florida
  - Sean A. Simon, MD, Miami, Florida
  - Pierini Esthetic Surgery, Miami, Florida
  - Imagos Plastic Surgery, Miami, Florida
  - Christopher Craft Cosmetic Surgery, Miami, Florida
  - Southeastern Plastic Surgery, Tallahassee, Florida
  - Dr. Joshua Halpern MD, PA, Tampa, Florida
  - The Swan Center for Plastic Surgery, Alpharetta, Georgia
  - Artisan Plastic Surgery, Atlanta, Georgia
  - North Atlanta Plastic Surgery, Atlanta, Georgia
  - Advanced Aesthetics, Fayetteville, Georgia
  - Marietta Plastic Surgery, Marietta, Georgia
  - Snodgrass and Robinson Plastic Surgery Specialists, Rome, Georgia
  - The Georgia Institute for Plastic Surgery, Savannah, Georgia
  - Barrington Plastic Surgery, Inverness, Illinois
  - MAE Plastic Surgery, Northbrook, Illinois
  - A New You Plastic Surgery & Laser Center, Oak Lawn, Illinois
  - Iowa Plastic Surgery, Davenport, Iowa
  - AMAE Plastic & Reconstructive Surgery, Birmingham, Michigan
  - Ellen A. Janetzke, MD, Bloomfield, Michigan
  - Partners in Plastic Surgery, Grand Rapids, Michigan
  - The Center for You, Traverse City, Michigan
  - Spa Renaissance & Renaissance Plastic Surgery, Troy, Michigan
  - Danielle DeLuca-Pytell, MD, PC, Troy, Michigan
  - Gryskiewicz Twin Cities Cosmetic Surgery, Burnsville, Minnesota
  - Parkcrest Plastic Surgery, St Louis, Missouri
  - Hankins and Sohn Plastic Surgery, Henderson, Nevada
  - Atlantic Plastic Surgery, Portsmouth, New Hampshire
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Doctors Plastic Surgery, Long Island City, New York
  - Piedmont Plastic Surgery & Dermatology - Blakeney, Charlotte, North Carolina
  - Providence Plastic Surgery & Skin Center, Charlotte, North Carolina
  - Piedmont Plastic Surgery & Dermatology - Cox Road, Gastonia, North Carolina
  - Piedmont Plastic Surgery & Dermatology Center - New Hope, Gastonia, North Carolina
  - Piedmont Plastic Surgery & Dermatology - Hickory, Hickory, North Carolina
  - Forsyth Plastic Surgery, Winston-Salem, North Carolina
  - Advanced Surgical Arts Center, Bismarck, North Dakota
  - The Columbus Institute for Plastic Surgery, Columbus, Ohio
  - Carp Cosmetic Surgery, Uniontown, Ohio
  - Tim R. Love, M.D., P.C., Oklahoma City, Oklahoma
  - Paul Glat, MD, PC, Bala-Cynwyd, Pennsylvania
  - Upstate Plastic Surgery, Greer, South Carolina
  - The Center for Dermatology and Plastic Surgery, Alcoa, Tennessee
  - Plastic Surgery Group, Chattanooga, Tennessee
  - Music City Plastic Surgery, Nashville, Tennessee
  - Ciaravino Plastic Surgery, Houston, Texas
  - Premier Plastic Surgery, Draper, Utah
  - Michael D. Marion Plastic Surgery, Lehi, Utah
  - Plastic Surgery of Fredericksburg, Fredericksburg, Virginia
  - Plastic Surgery Center of Hampton Roads, Newport News, Virginia
  - The Hague Center for Cosmetic and Plastic Surgery, Norfolk, Virginia
  - Richmond Plastic Surgeons, Richmond, Virginia
  - Kai Morimoto MD PLLC, Spokane Valley, Washington

IPD SHARING:
Plan to Share IPD: No